CLINICAL TRIAL: NCT06090487
Title: Is Sacubitril-valsartan Superior to Dapagliflozin in Improving Myocardial Function and Performance in Patients with Ischemic Cardiomyopathy Undergoing Coronary Artery Bypass Grafting Post-operatively in the Intensive Care Unit
Brief Title: Is Sacubitril-valsartan Superior to Dapagliflozin in Improving Myocardial Function Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Amr Gaber, lecturer clinical doctor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CABG
Record Dates: First submitted 2023-10-09; First posted 2023-10-19 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2023-10

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group sacubitril: (study group) (Other): This group includes (15) patients who will have 200 mg twice daily oral (5) sacubitril-valsartan 1 month before the operation.
  Interventions: Diagnostic Test: myocardial function after surgery
- Group dapagliflozin: (control group): (Other): This group includes (15) patients who will have a 10 mg single oral dose (4) 1 month before the operation.
  Interventions: Diagnostic Test: myocardial function after surgery

INTERVENTIONS:
Diagnostic Test: myocardial function after surgery — This group includes (15) patients who will have 200 mg twice daily oral (5) sacubitril-valsartan 1 month before the operation. transthoracic echo will be done before and after surgery, also total dose if inoptropic drugs will be noted

SUMMARY:
The aim of this study is to assess whether sacubitril-valsartan is more effective than dapagliflozin in improving function, myocardial performance in patients undergoing CABG operation or not

DETAILED DESCRIPTION:
Coronary revascularization has matured as a field since coronary artery bypass grafting (CABG) was first developed over 50 years ago, with diagnostic and treatment methods have advanced dramatically. CABG remains the standard of care for obstructive coronary artery disease, particularly for patients with multivessel disease or diabetes. (1) Despite significant therapeutic advances, patients with chronic heart failure (HF) remain at high risk for HF progression and death. Sacubitril/valsartan (previously known as LCZ696) is a first-in-class medicine that contains a neprilysin (NEP) inhibitor (sacubitril) and an angiotensin II (Ang-II) receptor blocker (valsartan). NEP is an endopeptidase that metabolizes different vasoactive peptides including natriuretic peptides, bradykinin and Ang-II. In consequence, its inhibition increases mainly the levels of both, natriuretic peptides (promoting diuresis, natriuresis and vasodilatation) and Ang-II whose effects are blocked by the angiotensin receptor blocker, valsartan (reducing vasoconstriction and aldosterone release). (2) Sacubitril-valsartan has been used selectively in patients undergoing coronary artery bypass grafting (CABG) and ischemic cardiomyopathy due to safety concerns. In a prospective observational study done by Narayan and his colleagues in Patients with Ischemic Cardiomyopathy Undergoing Off-Pump Coronary Artery Bypass Grafting Primary outcome was tolerability and safety profile. Thirty consecutive patients undergoing CABG with EF <40% were included. No mortality or readmissions occurred during 6 months' follow-up. One patient only experienced hypotension requiring discontinuation. Mild elevation in blood urea nitrogen, so Sacubitril-valsartan is well tolerated in patients with reduced EF undergoing CABG and proved its safety and efficacy. (3) Dapagliflozin is a highly potent, reversible and selective sodium-glucose cotransporter-2 inhibitor indicated worldwide for the treatment of type 2 diabetes. In numerous well-designed clinical studies dapagliflozin as monotherapy and combination therapy with other antihyperglycemic agents provided effective glycemic control and reduced bodyweight and blood pressure (BP) across a broad spectrum of patients. Dapagliflozin reduced the rate of cardiovascular (CV) death or hospitalization for heart failure (HF), did not adversely affect major adverse cardiovascular events (MACE) and possibly reduced progression of renal disease in patients with established atherosclerotic CV disease (CVD) or multiple risk factors for CVD. (4)

ELIGIBILITY:
Inclusion Criteria:

1. Age between 50 to 70 years old
2. DM type 2
3. ASA 3
4. Only 2 coronary grafts
5. Elective surgery
6. Bypass time less than 1 hour
7. Senior staff cardiothoracic

Exclusion Criteria:

1. ASA 4 or more
2. Emergency surgery
3. Bypass time of more than 1 hour
4. Coronary grafts of more than 2
5. Any allergy to the used drugs

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
heart rate | baseline just after the surgery and every 2 hours for 24 hours post operatively
  heart rate in beat per minute
Ejection fraction (EF) | 1.base line before start of medications 2.the day before surgery 3. just after surgery in the intensive care 4. 24 hours after surgery
  myocardial function using transthoracic echo
blood pressure | baseline just after the surgery then every 2 hours for 24 hours post operatively
  mean arterial blood pressure

SECONDARY OUTCOMES:
inotropic drugs | after addmitting to the intensive care just after surgery for the 1st 24 hours post operatively
  total dose of inotropic drugs

CONTACTS AND LOCATIONS:
Overall Officials: amr gaber, lecturer, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No